CLINICAL TRIAL: NCT01638728
Title: Change of Depth in a RAE Tube: Tube Fixation at the Midline or Angle and in a Neutral or Neck Extended Position
Status: Completed | Type: Observational
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Jong-Man Kang, Associate professor, Kyung Hee University Hospital at Gangdong
Other Study IDs: KHNMC 2012-039; KHNMC 039 (Other: KHNMC)
Record Dates: First submitted 2012-07-06; First posted 2012-07-12 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Depth of Tracheal Tube

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Endotracheal tube

SUMMARY:
The investigators compared the depth of the RAE tube [Preformed oral tracheal tubes were first described by Ring, Adair and Elwyn (therefore called RAE tubes)] when fixed at the midline and at the angle of the mouth, and after fixing the tube at the angle.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* Patients with anatomical defects of the face, neck, or upper airway

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients who are scheduled for elective surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
depth of tube | up to 1 hour
  from the tube tip to the carina

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea